CLINICAL TRIAL: NCT04618731
Title: Correlation Between Dental Caries Prevalence In Primary Teeth And First Permanent Molar of Children In Mixed Dentition Stage
Brief Title: Correlation Between Dental Caries Prevalence in Primary Teeth and First Permanent Moilar of Children in Mixed Dentition Stage
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nermeen Anwar Hamza, BDS, Cairo University
Other Study IDs: dental caries correlation
Record Dates: First submitted 2020-10-15; First posted 2020-11-06 (Actual); Last update posted 2020-11-06 (Actual); Status verified 2020-11

CONDITIONS: Dental Caries in Children
Keywords: risk factors, caries prediction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: caries prevalence def ,DMF — the examination will carried out on dental chair using diagnostic set

SUMMARY:
to find the clinical relation between caries experience in primary teeth and first permanent molar in mixed dentition stage using def index for primary teeth , DMF index for first permanent molars and to find the clinical relation between caries prevalence in the selected children in relation with other associated factors such as age, sex tooth brushing frequency, dietary habits and mother's attitude toward child's oral health.

DETAILED DESCRIPTION:
the problem for which the study held is lacking of data about relation between prevalence of dental caries in primary teeth and first permanent molar of the same child in mixed dentition stage, incidence of dental caries is influenced by number of risk factors such as age, sex dietary and oral hygiene habits identifying high risk individuals helps development of systemic approaches for preventive oral care programs world wide Dental caries is the major public health problem in most high income countries, affecting 60-90%of school children and the vast majority of adults. it also the most prevalent oral disease in several Asian and Latin American countries Although for the moment it appears to be less common and less severe in the greater part of Africa, the WHO report 2003 anticipates that in light of changing living conditions and dietary habits, the incidence of dental caries will increase in many of that continent's low income countries(WHO,2006)

ELIGIBILITY:
Inclusion Criteria:

* egyptian children
* children without systemic disease syndromes and disabilities
* first permanent molars fully erupted and in occlusion
* acceptance of the children's parents to participate in the study

Exclusion Criteria:

* any of first permanent molars aren't fully erupted or not in occlusion
* children suffering from any systematic disease that affect teeth development

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: children are selected from from children attending the diagnosis clinic of Department of pediatric dentistry and Dental public health
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
prevalence of dental caries in mixed dentition | baseline
  def(decayed primary tooth,decayed indicated for extraction tooth or filled primary tooth), DMF (decayed permanent tooth, missed of permanent tooth due to caries or filled permanent tooth) lower scores means better outcome
relation between caries prevalence and other associated factors | baseline
  answers of questionnaire

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Jokic NI, Bakarcic D, Jankovic S, Malatestinic G, Dabo J, Majstorovic M, Vuksan V. Dental caries experience in Croatian school children in Primorsko-Goranska county. Cent Eur J Public Health. 2013 Mar;21(1):39-42. doi: 10.21101/cejph.a3752. PMID 23741899
- [Result] Abbass MMS, Mahmoud SA, El Moshy S, Rady D, AbuBakr N, Radwan IA, Ahmed A, Abdou A, Al Jawaldeh A. The prevalence of dental caries among Egyptian children and adolescences and its association with age, socioeconomic status, dietary habits and other risk factors. A cross-sectional study. F1000Res. 2019 Jan 3;8:8. doi: 10.12688/f1000research.17047.1. eCollection 2019. PMID 30854195
- [Result] Albino J, Tiwari T. Preventing Childhood Caries: A Review of Recent Behavioral Research. J Dent Res. 2016 Jan;95(1):35-42. doi: 10.1177/0022034515609034. Epub 2015 Oct 5. PMID 26438210
- [Result] Doichinova L, Bakardjiev P, Peneva M. Assessment of food habits in children aged 6-12 years and the risk of caries. Biotechnol Biotechnol Equip. 2015 Jan 2;29(1):200-204. doi: 10.1080/13102818.2014.989180. Epub 2014 Dec 12. PMID 26019634